CLINICAL TRIAL: NCT01300247
Title: An Open-Label, Multicenter, Phase Ib Trial of GA101 (RO5072759) in Combination With Chemotherapy in Patients With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: A Study of Obinutuzumab (GA101; RO5072759) in Combination With Chemotherapy in Participants With Previously Untreated Chronic Lymphocytic Leukemia (CLL) (GALTON)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAO4779g; GO01298 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-02-14; First posted 2011-02-21 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; obinutuzumab; Bendamustine Hydrochloride; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obinutuzumab + Fludarabine + Cyclophosphamide (Experimental): Participants will receive 6 cycles (each 28-day cycle) of obinutuzumab (1000 mg IV infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycles 2-6), fludarabine (25 mg/m^2 IV, on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2-6), and cyclophosphamide (250 mg/m^2 IV on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2-6).
  Interventions: Drug: Fludarabine; Drug: Obinutuzumab; Drug: Cyclophosphamide
- Obinutuzumab + Bendamustine (Experimental): Participants will receive 6 cycles (each 28-day cycle) of obinutuzumab (1000 mg IV infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycles 2-6) and bendamustine (90 mg/m^2 IV, on Days 2 and 3 of Cycle 1 and Days 1 and 2 of Cycles 2-6).
  Interventions: Drug: Obinutuzumab; Drug: Bendamustine

INTERVENTIONS:
Drug: Fludarabine — Participants will receive 6 cycles (each 28-day cycle) of fludarabine at dose of 25 mg/m^2 IV, on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2-6.
  Arms: Obinutuzumab + Fludarabine + Cyclophosphamide
Drug: Obinutuzumab — Participants will receive 6 cycles (each 28-day cycle) of obinutuzumab at dose of 1000 mg IV infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycles 2-6.
  Other Names: RO5072759; GA101
Drug: Bendamustine — Participants will receive 6 cycles (each 28-day cycle) of bendamustine at dose of 90 mg/m^2 IV, on Days 2 and 3 of Cycle 1 and Days 1 and 2 of Cycles 2-6.
  Arms: Obinutuzumab + Bendamustine
Drug: Cyclophosphamide — Participants will receive 6 cycles (each 28-day cycle) of cyclophosphamide at dose of 250 mg/m^2 IV on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2-6.
  Arms: Obinutuzumab + Fludarabine + Cyclophosphamide

SUMMARY:
This open-label, 2-arm, nonrandomized, multicenter, Phase Ib study will investigate the safety and efficacy of obinutuzumab (RO5072759; GA101) administered in combination with chemotherapy (bendamustine or fludarabine + cyclophosphamide [FC] regimens) in participants with previously untreated cluster of differentiation 20 (CD20)-positive B-CLL. Participants will be enrolled to receive a maximum of 6 cycles of obinutuzumab (1000 milligrams [mg] intravenous [IV] infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycles 2 - 6) plus bendamustine (90 milligrams per meter square [mg/m^2] IV, on Days 2 and 3 of Cycle 1 and Days 1 and 2 of Cycles 2 - 6) on 28 day cycles or a maximum of 6 cycles of obinutuzumab (1000 mg IV infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycles 2 - 6) plus FC (fludarabine 25 mg/m^2 IV on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2 - 6; cyclophosphamide 250 mg/m^2 IV on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2 - 6) on 28 day cycles.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CD20-positive B-CLL
* Rai Stage III/IV or Binet Stage C disease
* Rai Stage I/II or Binet Stage B disease that requires treatment
* Adequate baseline bone marrow function, unless there is clear evidence of extensive bone marrow involvement with tumor infiltration, myelodysplasia, or hypocellularity
* No previous treatment for CLL by chemotherapy, radiotherapy, or immunotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of greater than (>) 6 months

Exclusion Criteria:

* Treatment with any other investigational agent or participation in another clinical trial within 28 days prior to the start of Cycle 1
* Transformation of CLL to aggressive B-cell malignancy
* Creatinine clearance less than equal to (<=) 60 milliliters per minute (mL/min), calculated according to the formula of Cockcroft and Gault
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2.5 times the upper limit of normal (ULN)
* Total bilirubin greater than equal to (>=) 3 x ULN
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* History of sensitivity to mannitol (if bendamustine is to be administered)
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease or pulmonary disease
* Known active bacterial, viral, fungal, mycobacterial, or other infection (excluding fungal infections of nail beds) or any major episode of infection requiring treatment with IV antibiotics or hospitalization (related to the completion of the course of antibiotics) within 4 weeks before the start of Cycle 1
* Recent major surgery (within 4 weeks prior to the start of Cycle 1), other than for diagnosis
* Known infection with human immunodeficiency virus (HIV) seropositive status
* Presence of positive test results for hepatitis B (hepatitis B virus [HBV] surface antigen [HBsAg] and/or total hepatitis B core antibody [anti-HBc]) or hepatitis C (hepatitis C virus [HCV] antibody serology testing). Participants with chronic HBV infection, occult HBV infection, or past HBV infection will be excluded. Participants who have received IV immunoglobulin within 3 months of enrollment and who are anti-HBc positive but HBV deoxyribonucleic acid (DNA) negative will be considered for inclusion on the study by the Medical Monitor on a case-by-case basis. Participants positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA).
* Women who are pregnant or lactating
* Fertile men or women of childbearing potential unless 1) surgically sterile or 2) using an adequate measure of contraception such as oral contraceptives, intrauterine device, or barrier method of contraception in conjunction with spermicidal jelly
* Concurrent (or within 7 days prior to the first dose of study treatment) systemic corticosteroid use except low-dose corticosteroid therapy used to treat an illness other than lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (18):
- United States (18):
  - Huntsville, Alabama
  - Duarte, California
  - La Jolla, California
  - Los Angeles, California
  - Southington, Connecticut
  - Tampa, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Boston, Maryland
  - Boston, Massachusetts
  - Saint Louis Park, Minnesota
  - Springfield, Missouri
  - Rochester, New York
  - Houston, Texas
  - Seattle, Washington
  - Tacoma, Washington
  - Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown JR, O'Brien S, Kingsley CD, Eradat H, Pagel JM, Lymp J, Hirata J, Kipps TJ. Obinutuzumab plus fludarabine/cyclophosphamide or bendamustine in the initial therapy of CLL patients: the phase 1b GALTON trial. Blood. 2015 Apr 30;125(18):2779-85. doi: 10.1182/blood-2014-12-613570. Epub 2015 Mar 13. PMID 25769620

RESULTS

PARTICIPANT FLOW:
Groups:
- Obinutuzumab + Fludarabine + Cyclophosphamide: Participants received 6 cycles (each 28-day cycle) of obinutuzumab (1000 milligrams [mg] intravenous [IV] infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycles 2-6), fludarabine (25 milligrams per meter square [mg/m^2] IV, on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2-6) and cyclophosphamide 250 mg/m^2 IV on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2-6). The Cycle 1 Day 1 dose of obinutuzumab was split over two days (Cycle 1 Day 1 and Cycle 1 Day 2).
- Obinutuzumab + Bendamustine: Participants received 6 cycles (each 28-day cycle) of obinutuzumab (1000 mg IV infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycles 2-6) and bendamustine (90 mg/m^2 IV, on Days 2 and 3 of Cycle 1 and Days 1 and 2 of Cycles 2-6).
Period: Overall Study
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Started | 21 | 20
Completed | 17 | 18
Not Completed | 4 | 2
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Non-Compliance | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety-Evaluable population included all participants who received any amount of study treatment.
Groups:
- Obinutuzumab + Fludarabine + Cyclophosphamide: Participants received 6 cycles (each 28-day cycle) of obinutuzumab (1000 mg IV infusion, on Days 1, 8 and 15 of Cycle 1 and Day 1 of Cycles 2-6), fludarabine (25 mg/m^2 IV, on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2-6) and cyclophosphamide 250 mg/m^2 IV on Days 2, 3 and 4 of Cycle 1 and Days 1, 2 and 3 of Cycles 2-6). The Cycle 1 Day 1 dose of obinutuzumab was split over two days (Cycle 1 Day 1 and Cycle 1 Day 2).
- Total: Total of all reporting groups
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (11.1) | 62.0 (9.0) | 59.8 (10.2)
Gender [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Human Anti-Human Antibodies (HAHAs)
Time Frame: Cycle 1 Day 1 (cycle length = 28 days) up to clinical data cutoff date 24 January 2013 (up to approximately 1.75 years)
Population: Safety evaluable population
Measure: Number; unit: participants
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 21 | 20
participants | 0 | 0

2. Secondary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) of Obinutuzumab
Description: AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: Pre-dose on Cycle (C) 1 Day (D) 1, immediately after end of infusion (0.5 hour), 0.5 hour of split dose of C1D2, pre-dose and immediately after end of infusion on C1D3, 8, 15, C2D1, C4D1, C6D1 and at progression (up to 1.75 year overall)
Population: The pharmacokinetic (PK) variables could not be calculated as the PK samples were not collected accurately.
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Obinutuzumab
Time Frame: as for outcome 2
Population: The PK variables could not be calculated as the PK samples were not collected accurately.
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Trough Plasma Concentration (Ctrough) of Obinutuzumab
Time Frame: Pre-dose on C1D1, C1D3, 8, 15, C2D1, C4D1, C6D1
Population: The PK variables could not be calculated as the PK samples were not collected accurately.
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Clearance of Obinutuzumab
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population PK modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Pre-dose on C1D1, immediately after end of infusion (0.5 hour), 0.5 hour of split dose of C1D2, pre-dose and immediately after end of infusion on C1D3, 8, 15, C2D1, C4D1, C6D1 and at progression (up to 1.75 year overall)
Population: The PK variables could not be calculated as the PK samples were not collected accurately.
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Volume of Distribution of Obinutuzumab
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: as for outcome 2
Population: The PK variables could not be calculated as the PK samples were not collected accurately.
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Half-Life of Obinutuzumab
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 2
Population: The PK variables could not be calculated as the PK samples were not collected accurately.
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants With Objective Response, Assessed According to International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Guidelines
Description: Objective response was defined as a complete response (CR), CR with incomplete marrow recovery (CRi) or partial response (PR), as determined by investigator. CR:required peripheral blood lymphocytes <4x10^9/L; absence of lymphadenopathy; no hepatomegaly or splenomegaly by physical examination as determined by measurement below relevant costal margin; absence of disease/constitutional symptoms; bone marrow at least normocellular for age, with <30% of nucleated cells being lymphocytes. PR:Greater than equal to (>=) 50% decrease in peripheral blood lymphocyte count, >=50% reduction in lymphadenopathy, >=50% reduction of liver and/or spleen enlargement, either neutrophil, platelet, or hemoglobin (Hb) recovery. CRi:met all CR criteria including confirmed lymphocyte infiltration <30%; may not meet Hb, platelet or neutrophil count recovery. The 95% confidence interval (CI) was estimated by Clopper-Pearson method. The end of treatment response visit occurred 2-3 months after end of treatment.
Time Frame: Baseline up to relapse or progression or death from any cause, whichever occurred first up to end of treatment response visit (up to approximately 9 months)
Population: Safety evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 21 | 20
percentage of participants | 61.9 [38.44 to 81.89] | 90.0 [68.30 to 98.77]

9. Secondary Outcome: Duration of Objective Response (DOR), Assessed by the Investigator According to IWCLL Guidelines
Description: DOR for participants with OR: time from first CR, CRi or PR to disease progression (DP), relapse, or death, assessed by the investigator. DP: >=50% increase in lymphocytes to at least 5x10^9/L;new palpable lymph nodes (>15 millimeters [mm] in longest diameter) or any new extra-nodal lesion; >=50% increase in the longest diameter of any previous site of lymphadenopathy; >=50% increase in the enlargement of the liver and/or spleen; transformation to a more aggressive histology. CR:peripheral blood lymphocytes (PBL) <4x10^9/L; no lymphadenopathy; no hepatomegaly or splenomegaly (below relevant costal margin); no symptoms; bone marrow at least normocellular for age, with <30% of nucleated cells being lymphocytes. PR: >=50% decrease in PBL, >=50% reduction in lymphadenopathy, >=50% reduction of liver and/or spleen enlargement, either neutrophil, platelet, or hemoglobin (Hb) recovery. CRi: met CR criteria, lymphocyte infiltration <30%; may not meet Hb, platelet or neutrophil count recovery.
Time Frame: From first documented objective response up to disease progression or relapse or death, whichever occurred first (up to approximately 6 months)
Population: Safety evaluable population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 21 | 20
percentage of participants | NA [NA to NA] — Not estimated as not enough data captured in this arm at 6 months | 100.00 [100.00 to 100.00]

10. Secondary Outcome: Percentage of Participants Who Were Alive and Progression Free
Description: Progressive disease assessed using IWCLL: >=50% increase in the absolute number of circulating lymphocytes to at least 5x10^9/L; Appearance of new palpable lymph nodes (>15 millimeters [mm] in longest diameter) or any new extra-nodal lesion; >=50% increase in the longest diameter of any previous site of lymphadenopathy; >=50% increase in the enlargement of the liver and/or spleen; transformation to a more aggressive histology.
Time Frame: Baseline up to relapse or progression or death from any cause, whichever occurred first, up to end of study (up to approximately 4 years)
Population: Safety evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 21 | 20
percentage of participants | 90.5 | 90.0

11. Secondary Outcome: Percentage of Participants Who Were Alive
Time Frame: as for outcome 10
Population: Safety evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 21 | 20
percentage of participants | 95.2 | 95.0

12. Secondary Outcome: Percentage of Participants Who Had B-Cell Depletion
Description: B-cell depletion was defined as cluster of differentiation 19 (CD19) <0.07×10^9/L and could occur only after at least one dose of study drug had been administered.
Time Frame: Up to the end of the treatment period, and follow-up at 6 months, 6-12 months and after 12 months up to end of study (up to approximately 4 years)
Population: Safety evaluable population
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 21 | 20
percentage of participants
  End of the treatment period | 90.5 | 100.0
  Follow-up at 6 months | 85.7 | 100.0
  Within 6-12 months of follow-up | 81.0 | 100.0
  After 12 months follow-up | 47.6 | 70.0

13. Secondary Outcome: Percentage of Participants Who Had B-Cell Recovery
Description: B-cell recovery was defined as CD19 >=0.07×10^9/L, where participants' CD19 were previously depleted. B-cell recovery was only considered possible when the participant had received the last dose of study treatment.
Time Frame: Follow-up at 6 months, 6-12 months and after 12 months up to end of study (up to approximately 4 years)
Population: Safety evaluable population
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 21 | 20
percentage of participants
  Follow-up at 6 months | 0 | 0
  Within 6-12 months of follow-up | 9.5 | 0
  After 12 months follow-up | 42.9 | 30.0

ADVERSE EVENTS:
Time Frame: Up to the end of the study (up to approximately 4 years).
Description: All adverse events (related and unrelated to treatment) were to be collected up to 28 days after the last dose of obinutuzumab. After 28 days after the last dose of obinutuzumab, investigators were to report only serious adverse events that were attributed to obinutuzumab; these were to be reported to Genentech/Roche Drug Safety indefinitely (even if the study was closed). Significant abnormalities in laboratory parameters were reported as adverse events.
Arm/Group | Obinutuzumab + Fludarabine + Cyclophosphamide | Obinutuzumab + Bendamustine
Serious Adverse Events (participants affected / at risk) | 6/21 | 11/20
Other Adverse Events (participants affected / at risk) | 21/21 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + Fludarabine + Cyclophosphamide (N=21) | Obinutuzumab + Bendamustine (N=20)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 3
Tachycardia (Cardiac disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + Fludarabine + Cyclophosphamide (N=21) | Obinutuzumab + Bendamustine (N=20)
Neutropenia (Blood and lymphatic system disorders) | 5 | 10
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Cytopenia (Blood and lymphatic system disorders) | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 16 | 12
Constipation (Gastrointestinal disorders) | 10 | 7
Vomiting (Gastrointestinal disorders) | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 10
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Epigastric discomfort (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 12 | 7
Pyrexia (General disorders) | 5 | 8
Chills (General disorders) | 2 | 7
Oedema peripheral (General disorders) | 2 | 1
Pain (General disorders) | 0 | 3
Asthenia (General disorders) | 1 | 1
Injection site pain (General disorders) | 0 | 2
Axillary pain (General disorders) | 0 | 1
Catheter site pain (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Sinusitis (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 1
Candida infection (Infections and infestations) | 2 | 0
Paronychia (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 2 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 5
Headache (Nervous system disorders) | 0 | 5
Memory impairment (Nervous system disorders) | 0 | 2
Aphonia (Nervous system disorders) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Restless leg syndrome (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 3
Anxiety (Psychiatric disorders) | 0 | 5
Communication disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus generalized (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Butterfly rash (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 4
Hypotension (Vascular disorders) | 1 | 2
Phlebitis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1
Phlebitis superficial (Vascular disorders) | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 16 | 11
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Radiotherapy (Surgical and medical procedures) | 0 | 1
Sinus operation (Surgical and medical procedures) | 0 | 1

LIMITATIONS AND CAVEATS:
The interim data reported here (up to clinical cutoff date of 24 January 2013) were for participants who had completed treatment response assessment, which took place approximately 2 months after the last infusion of study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.